CLINICAL TRIAL: NCT03424434
Title: Underreporting of Occupational Blood Exposure (OBE) Among Medical Staff at an University Hospital Center (UHC) in 2017
Brief Title: Underreporting of Occupational Blood Exposure (OBE) Among Medical Staff at an University Hospital Center (UHC) in 2017 (OBE PRACTITIONERS UHC 2017)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0883
Record Dates: First submitted 2018-01-23; First posted 2018-02-07 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-03

CONDITIONS: Health Professional
Keywords: Occupational blood exposure; underreporting; medical; hospital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical staff of an UHC, practitioners and residents: The target population is practitioners and residents who works at hospital in an UHC, they are also specialists, surgeons, dental surgeons.
  Interventions: Other: Survey diffusion

INTERVENTIONS:
Other: Survey diffusion — The study consists in a survey diffusion during several weeks by emailing each practitioner and resident and inviting them to participate to a questionnaire about occupational blood exposure. This survey is strictly anonymous. No identity data is required, only age, gender, function, surgical or medical specialty, work quota and hospital group they belong. This survey is diffused in four UHC (Lyon, Grenoble, Clermont-Ferrand and Saint-Etienne) in France.

SUMMARY:
Regarding 30 to 50% of occupational blood exposure (OBE) are underreporting among health professionals, it's to highlight that the part of medical professionals in OBE reporting is among the lowest (1996 to 2016). The current study is aiming to evaluate the underreporting of this specific occupational accident among medical staff for the year 2017. The investigators are supposing this is declining and the part of OBE reporting is better than before. So the current situation concerning OBE underreporting for medical staff in an University Hospital Center (UHC), 20 years after the first study, is our main purpose.

ELIGIBILITY:
Inclusion Criteria:

* Any medical or surgical health professional
* practitioner and resident
* working in an UHC
* without distinction of medical or surgical specialty
* having a professional mailbox

Exclusion Criteria:

* All paramedical health professionals (example: nurses) and pharmacists
* Any medical or surgical health professional working full-time outside an UHC
* Any medical or surgical health professional with exclusive liberal activity outside an UHC
* Administrative and technical staff of an UHC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University Hospital Center (UHC) Medical staff
Sampling Method: Non-Probability Sample
Enrollment: 1493 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-05-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of underreporting occupational blood exposure (OBE) among the medical staff at an University Hospital Center (UHC) for the year 2017 | 1 day
  This evaluation consists in collecting, during the diffusion of a survey, the number of OBE the medical professional is victim of and the number of OBE is reported to deduce the number of non-reported OBE, over the period of interest which is the year 2017.

SECONDARY OUTCOMES:
The occurrence circumstances of OBE | 1 day
  These questions are gathered in a table and concern different sorts of contaminated needlesticks, blood projections, cut or wound and the positive serologic status for the source patient.
  This specific outcome is qualitatively evaluated with questions relating to the occurence circumstances of OBE with a choice of standards answers (Yes, always - Often - Sometimes - No, never).
The part of each factor, related to the professional activity and to the OBE itself, in the OBE reporting. | 1 day
  Some questions are gathered in a table and propose 15 differents reasons that can condition the OBE reporting, such as lack of time, fear of judgment, repetition of OBE, unknowing of reporting procedure, lack of standards precautions, only antisepsis maneuvers sufficient, source patient considered as safe, procedure to report considered complex, fear of career consequences, lack of witness, night work, negatives serologies for the source patient, fear of the serological follow-up, fear observing an antiretroviral treatment, ignorance that an OBE was a true one. For each factor, a percentage will be measured as indicative of its importance in the OBE underreporting.
  This specific outcome considering various factors that can influence the reporting of an OBE is evaluated by several questions with a yes or no answer.
Involvement of behaviors of underreporting medical professionals | 1 day
  Using two tables, several measures recommanded about the biological risk in hospital environment (including OBE) are discussed. These differents measures are considered as primary and secondary preventive behaviors. For each measure, we examine its frequency as indicative of its implication in the OBE underreporting.
  This outcome is evaluated with questions on vaccination, immunization, wearing of personal protective equipment and realization of the antisepsis maneuvers, realization of serologies for source patient and personal ones, with a choice of standards answers (Yes, always - Often - Sometimes - No, never).
Practitioners knowledges about the specific infectious risk of OBE | 1 day
  On a first table, the participant has to choose one of the four rates proposed (30% - 1 to 3% - 0,3% - < 0,3%) to evaluate the risk of seroconversion after percutaneous contact with infected blood by HIV or hepatitis B virus (HBV) or hepatitis C virus (HCV). On a second table, the participant has to choose a time limit (Immediately - within 4 hours - within 48 hours - up to 7 days) for different situations near OBE occurence, it concerns antisepsis maneuvers, prophylactic antiretroviral treatment, initial personal serological status and source patient serological status.
  A test is proposed to evaluate knowledges about the infectious risk related to OBE, this test is optional, grouping together seven simple choice questions.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble Alpes, La Tronche
  - Groupement Hospitalier Sud, Pierre-Bénite
  - CHU de Saint-Etienne, Saint-Etienne